CLINICAL TRIAL: NCT04167982
Title: Efficacy and Safety of Painless 5-aminolevulinic Acid Photodynamic Therapy for the Treatment of Moderate and Severe Acne Vulgaris-- A Multi-center, Randomized Controlled Clinical Trial
Brief Title: Efficacy and Safety of Painless 5-aminolevulinic Acid Photodynamic Therapy for Moderate and Severe Acne Vulgaris
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Dermatology Hospital (Other)
Collaborators: Huadong Hospital (Other); RenJi Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2019-11
Record Dates: First submitted 2019-10-26; First posted 2019-11-19 (Actual); Last update posted 2020-11-24 (Actual); Status verified 2020-11

CONDITIONS: Acne
Keywords: Acne; low-dose isotretinoin; Photodynamic Therapy; Painless
MeSH Terms: conditions — Acne Vulgaris | interventions — Isotretinoin

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Painless Photodynamic Therapy(P-PDT) group (Experimental): The painless photodynamic therapy group underwent narrow-band light-emitting diode (LED) irradiation (630 nm; 150 J/cm2) after applying 5% 5-aminolevulinic acid(ALA) cream for 30min. A repeat treatment was administered once weekly for a maximum of 5 times. Blood samples, urine routine, blood biochemistry and electrocardiogram were performed before treatment and after treatment.
  Interventions: Procedure: Aminolevulinic acid photodynamic therapy
- conventional-dose isotretinoin group (Active Comparator): Patients in the conventional-dose isotretinoin group were given oral isotretinoin 0.5 mg/kg daily for 6 months, and the cumulative dose was 90 mg/kg. Time for subsequent visit: once every two weeks during the 1st and 2nd months, monthly during 3rd to 6th months. Blood samples, urine routine, blood biochemistry and electrocardiogram were performed before treatment and 2nd , 6th months after treatment.
  Interventions: Drug: Oral conventional-dose isotretinoin
- low-dose isotretinoin group (Active Comparator): Patients in the low-dose isotretinoin group were given oral isotretinoin 0.2 mg/kg daily for 6 months, and the cumulative dose was 36 mg/kg. Time for subsequent visit: once every two weeks during the 1st and 2nd months, monthly during 3rd to 6th months. Blood samples, urine routine, blood biochemistry and electrocardiogram were performed before treatment and 2nd , 6th months after treatment.
  Interventions: Drug: Oral low-dose isotretinoin

INTERVENTIONS:
Procedure: Aminolevulinic acid photodynamic therapy — Aminolevulinic acid photodynamic therapy
  Arms: Painless Photodynamic Therapy(P-PDT) group
Drug: Oral conventional-dose isotretinoin — Conventional-dose isotretinoin
  Arms: conventional-dose isotretinoin group
Drug: Oral low-dose isotretinoin — low-dose isotretinoin
  Arms: low-dose isotretinoin group

SUMMARY:
This study is being done to compare a new, continuous illumination and short Incubation time regimen of 5-aminolevulinic acid photodynamic therapy (painless ALA- PDT) to low-dose and conventional dose of oral isotretinoin for treatment of moderate or severe acne vulgaris. The hypothesis is that the painless ALA- PDT will be equally or more efficacious as oral isotretinoin, and taking effect more quickly with less adverse effect.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosed with moderate to severe acne
* Male and female patients of age between 18-40 years old
* All patients read the instructions of the subject, willing to follow the program requirements
* No other topical treatment received within 2 weeks prior to enrollment
* No systemic treatment was given within 4 weeks prior to enrollment
* Patients were unsuitable for other treatments for various reasons and signed informed consent when they had informed other alternatives and agreed to take pictures of the lesion

Exclusion Criteria:

* Those who did not complete the informed consent
* The lesions belongs to any of the following conditions: There is damage and inflammation, which may lead to the drug entering the open wound
* Patients with skin photoallergic diseases, porphyria
* Known to have a history of allergies to test drugs (porphyrins) and their chemically similar drugs
* Patients with other obvious diseases that may affect the evaluation of efficacy
* Scars or patients with a tendency to form scars
* Known to have severe immune dysfunction, or long-term use of glucocorticoids and immunosuppressants
* Severe heart, liver, kidney disease; with hereditary or acquired coagulopathy
* Those with severe neurological, psychiatric or endocrine diseases
* Women who are pregnant, breast-feeding or using inappropriate contraceptives -Those with a history of drug abuse; those who have participated in other drug clinical trials within 4 weeks before treatment

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 234 (Estimated)
Dates: Start 2020-03-28 (Actual); Primary Completion 2022-11-30 (Estimated); Study Completion 2022-11-30 (Estimated)

PRIMARY OUTCOMES:
The clearance rate of Moderate or Severe Acne | The clearance rate of Moderate or Severe Acne will be measured at 1st month after the last treatment
  The clearance rate of Moderate or Severe Acne will be measured at 1st month after the last treatment

SECONDARY OUTCOMES:
Pain assessment | immediately, 1st minute, 3rd minute, 5th minute, 7th minute, 10th minute and 2nd hour, 12th hour, 24th hour and 48th hour after treatment
  The pain will be assessed using Visual Analogue Scale (NRS) with a score range of 0-10. The higher the score, the greater the pain, with 0 being no pain and 10 being the most unbearable pain. Pain will be measured at different time points during and after every treatment (including immediately, 1st minute, 3rd minute, 5th minute, 7th minute, 10th minute and 2nd hour, 12th hour, 24th hour and 48th hour after treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Xiuli Wang, MD PhD, Study Chair — Shanghai Skin Disease Hospital
Locations (1):
- Lei Shi, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: CSR
Time Frame: One year after finishing this study and for permanency
Access Criteria: anyone who search pubmed